CLINICAL TRIAL: NCT04396535
Title: Randomized Phase II Study of Standard Chemotherapy With Docetaxel With or Without Bintrafusp Alfa in Patients With Advanced NSCLC After Progressing on a Combination of Anti-PD-1/PD-L1 Agents and Chemotherapy
Brief Title: Docetaxel With or Without Bintrafusp Alfa for the Treatment of Advanced Non-small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: EMD Serono recommendation based on three other studies that failed to show benefit for bintrafusp alfa
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MC1821; NCI-2020-02975 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1821 (Other: Mayo Clinic in Rochester); 19-010887 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2020-05-14; First posted 2020-05-20 (Actual); Results first posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2024-01

CONDITIONS: Advanced Lung Non-Small Cell Carcinoma; Stage III Lung Cancer AJCC v8; Stage IIIA Lung Cancer AJCC v8; Stage IIIB Lung Cancer AJCC v8; Stage IIIC Lung Cancer AJCC v8; Stage IV Lung Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8
MeSH Terms: conditions — Lung Neoplasms | interventions — bintrafusp alfa protein, human; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (docetaxel, bintrafusp alfa) (Experimental): Patients receive docetaxel IV over 1 hour and bintrafusp alfa IV over 60 minutes on day 1. Treatment repeats every 3 weeks for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive bintrafusp alfa IV over 60 minutes on day 1. Cycles repeat every 3 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bintrafusp Alfa; Drug: Docetaxel
- Arm II (docetaxel) (Active Comparator): Patients receive docetaxel IV over 1 hour on day 1. Cycles repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. Patients who experience disease progression may crossover to Arm I and receive bintrafusp alfa alone.
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Bintrafusp Alfa — Given IV
  Other Names: Anti-PDL1/TGFb Trap MSB0011359C; M7824; MSB0011359C
  Arms: Arm I (docetaxel, bintrafusp alfa)
Drug: Docetaxel — Given IV
  Other Names: Docecad; RP56976; Taxotere; Taxotere Injection Concentrate

SUMMARY:
This phase II trial studies how well docetaxel works with or without bintrafusp alfa in treating patients with non-small cell lung cancer that has spread to other places in the body (advanced). Chemotherapy drugs, such as docetaxel, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Immunotherapy with bintrafusp alfa, may induce changes in body's immune system and may interfere with the ability of tumor cells to grow and spread. Giving docetaxel and bintrafusp alfa in combination may work better in treating non small-cell lung cancer compared to docetaxel alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the progression-free survival (PFS) of bintrafusp alfa in combination with docetaxel versus (vs) docetaxel alone.

SECONDARY OBJECTIVES:

I. To evaluate overall survival of bintrafusp alfa in combination with docetaxel vs docetaxel alone.

II. To evaluate overall response rates of bintrafusp alfa in combination with docetaxel vs docetaxel alone.

III. To evaluate duration of response of bintrafusp alfa in combination with docetaxel vs docetaxel alone.

IV. To evaluate the safety of bintrafusp alfa in combination with docetaxel vs docetaxel alone.

CORRELATIVE RESEARCH OBJECTIVES:

I. To evaluate PD-L1, TGF-beta, and TMB as potential predictive markers of clinical response in tumor biopsies and in plasma.

II. To evaluate biomarkers associated with inhibition of TGF-beta and PD-L1. III. To evaluate the changes in immune system using mass cytometry in response to TGF-beta and PD-L1 inhibition.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive docetaxel intravenously (IV) over 1 hour and bintrafusp alfa IV over 60 minutes on day 1. Treatment repeats every 3 weeks for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive bintrafusp alfa IV over 60 minutes on day 1. Cycles repeat every 3 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive docetaxel IV over 1 hour on day 1. Cycles repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. Patients who experience disease progression may crossover to Arm I and receive bintrafusp alfa alone.

After completion of study treatment, patients are followed up at 30 days and then every 3 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Histological confirmation of non-small cell lung cancer (NSCLC) with advanced disease
* Prior treatment required:

  * Anti-PD1/PD-L1 agent in combination with platinum-based chemotherapy
* Measurable disease

  * NOTE: Tumor lesions in a previously irradiated area are not considered measurable disease; Disease that is measurable by physical examination only is not eligible
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* Hemoglobin >= 9.0 g/dL (obtained =< 14 days prior to registration)
* Absolute neutrophil count (ANC) >= 1500/mm^3 (obtained =< 14 days prior to registration)
* Platelet count >= 100,000/mm^3 (obtained =< 14 days prior to registration)
* Total bilirubin =< upper limit of normal (ULN) (obtained =< 14 days prior to registration)
* Alanine aminotransferase (ALT/serum glutamate pyruvate transaminase [SGPT]) and aspartate transaminase (AST/serum glutamic-oxaloacetic transaminase [SGOT]) =< 1.5 x ULN (obtained =< 14 days prior to registration)
* Alkaline phosphatase <= 2.5 x ULN (obtained =< 14 days prior to registration)
* Prothrombin time (PT)/international normalized ratio (INR)/activated partial thromboplastin time (aPTT) =< 1.5 x ULN OR if patient is receiving anticoagulant therapy INR or aPTT is within target range of therapy (obtained =< 14 days prior to registration)
* Calculated creatinine clearance >= 30 ml/min using the Cockcroft-Gault formula (obtained =< 14 days prior to registration)
* Negative pregnancy test done =< 7 days prior to registration, for persons of childbearing potential only

  * NOTE: If a urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Willing to use birth control as follows:

  * If able to become pregnant: Willing to use birth control during treatment and for 6 months after last dose of docetaxel and/or bintrafusp alfa, whichever is later
  * If able to father a child: Willing to use birth control with partners able to become pregnant during treatment and for 3 months after last dose of docetaxel and/or bintrafusp alfa, whichever is later
* Provide written informed consent
* Willingness to provide mandatory blood specimens for correlative research
* Willingness to provide mandatory tissue specimens for correlative research
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)
* CROSSOVER ELIGIBILITY: Documented disease progression =< 28 days prior to crossover registration
* CROSSOVER ELIGIBILITY: No contraindications to bintrafusp alfa at the time of crossover registration
* CROSSOVER ELIGIBILITY: Patient and physician agree to try crossover treatment with bintrafusp alfa
* CROSSOVER ELIGIBILITY: Provide written informed consent

Exclusion Criteria:

* Any of the following because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown:

  * Pregnant persons
  * Nursing persons
  * Persons of childbearing potential who are unwilling to employ adequate contraception
* Any of the following prior therapies:

  * Surgery =< 4 weeks prior to registration
  * Chemotherapy =< 4 weeks prior to registration
  * Received single agent anti-PD1/PD-L1 as first line therapy for metastatic disease
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Or psychiatric illness/social situations that would limit compliance with study requirements
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Other active malignancy =< 5 years prior to registration

  * EXCEPTIONS: Non-melanotic skin cancer or carcinoma-in-situ of the cervix

    * NOTE: If there is a history of prior malignancy, they must not be receiving other specific treatment for their cancer
* History of myocardial infarction =< 6 months, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* Known primary central nervous system (CNS) malignancy or symptomatic CNS metastases are excluded, with the following exceptions:

  * Patients with asymptomatic untreated CNS disease may be enrolled, provided all of the following criteria are met:

    * Evaluable or measurable disease outside the CNS
    * No metastases to brain stem, midbrain, pons, medulla, cerebellum, or within 10 mm of the optic apparatus (optic nerves and chiasm)
    * No history of intracranial hemorrhage or spinal cord hemorrhage
    * No ongoing requirement for dexamethasone for CNS disease; patients on a stable dose of anticonvulsants are permitted
    * No neurosurgical resection or brain biopsy =< 28 days prior to registration
  * Patients with asymptomatic treated CNS metastases may be enrolled, provided all the criteria listed above are met as well as the following:

    * Radiographic demonstration of improvement upon the completion of CNS-directed therapy and no evidence of interim progression between the completion of CNS-directed therapy and the screening radiographic study
    * No stereotactic radiation or whole-brain radiation =< 28 days prior to registration
    * Screening CNS radiographic study >= 4 weeks from completion of radiotherapy and >= 2 weeks from discontinuation of corticosteroids
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* History or current evidence of bleeding disorder, including bleeding diathesis, i.e., any hemorrhage/bleeding event of Common Terminology Criteria for Adverse Events (CTCAE) grade >= 2 in =< 28 days prior to registration
* Taking oral prednisone of >= 10 mg daily or equivalent
* Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis; cirrhosis; fatty liver; and inherited liver disease. Notes:

  * Patients with past or resolved hepatitis B infection (defined as having a negative hepatitis B surface antigen [HBsAg] test and a positive anti-HBc [antibody to hepatitis B core antigen] antibody test) are eligible
  * Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV ribonucleic acid (RNA)
* History or risk of autoimmune disease, including, but not limited to, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjogren's syndrome, Bell's palsy, Guillain-Barre syndrome, multiple sclerosis, autoimmune thyroid disease, vasculitis, or glomerulonephritis. Notes:

  * Patients with a history of autoimmune hypothyroidism on a stable dose of thyroid replacement hormone are eligible
  * Patients with controlled type 1 diabetes mellitus on a stable insulin regimen are eligible
  * Patients with eczema, psoriasis, lichen simplex chronicus of vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis would be excluded) are permitted provided that they meet the following conditions:

    * Patients with psoriasis must have a baseline ophthalmologic exam to rule out ocular manifestations
    * Rash must cover less than 10% of body surface area (BSA)
    * Disease is well controlled at baseline and only requiring low potency topical steroids (e.g., hydrocortisone 2.5%, hydrocortisone butyrate 0.1%, fluocinolone 0.01%, desonide 0.05%, alclometasone dipropionate 0.05%)
    * No acute exacerbations of underlying condition within the last 12 months (not requiring psoralen plus ultraviolet A radiation [PUVA], methotrexate, retinoids, biologic agents, oral calcineurin inhibitors; high potency or oral steroids)
* Known active human immunodeficiency virus (HIV) infection (defined as patients who are not on anti-retroviral treatment and have detectable viral load and CD4+ < 500/ml)

  * NOTE: HIV-positive patients who are well controlled on anti-retroviral therapy are allowed to enroll
* History of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis on screening chest computed tomography (CT) scan. Note: History of radiation pneumonitis in the radiation field (fibrosis) is permitted
* Severe infections =< 4 weeks prior to registration, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia
* History of peripheral neuropathy >= grade 2
* Known hypersensitivity to docetaxel or polysorbate 80

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-10-23 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Leventakos, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was projected to accrue 80 patients and only accrued 10 due to early termination of study.
Groups:
- Arm I (Docetaxel, Bintrafusp Alfa): Patients receive docetaxel IV over 1 hour and bintrafusp alfa IV over 60 minutes on day 1. Treatment repeats every 3 weeks for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive bintrafusp alfa IV over 60 minutes on day 1. Cycles repeat every 3 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity.> >>
  >
  >> Bintrafusp Alfa: Given IV>
  >>
  >
  >> Docetaxel: Given IV
- Arm II (Docetaxel): Patients receive docetaxel IV over 1 hour on day 1. Cycles repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. Patients who experience disease progression may crossover to Arm I and receive bintrafusp alfa alone.>
  >>
  >
  >> Docetaxel: Given IV
Period: Initial Study
Arm/Group | Arm I (Docetaxel, Bintrafusp Alfa) | Arm II (Docetaxel)
Started | 6 | 4
Completed | 6 | 3
Not Completed | 0 | 1
Period: Crossover
Arm/Group | Arm I (Docetaxel, Bintrafusp Alfa) | Arm II (Docetaxel)
Started | 0 | 1
Completed | 0 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm I (Docetaxel, Bintrafusp Alfa): Patients receive docetaxel IV over 1 hour and bintrafusp alfa IV over 60 minutes on day 1. Treatment repeats every 3 weeks for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive bintrafusp alfa IV over 60 minutes on day 1. Cycles repeat every 3 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity.>> >> Bintrafusp Alfa: Given IV>>
  >> Docetaxel: Given IV
- Arm II (Docetaxel): Patients receive docetaxel IV over 1 hour on day 1. Cycles repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. Patients who experience disease progression may crossover to Arm I and receive bintrafusp alfa alone.>>
  >> Docetaxel: Given IV
- Total: Total of all reporting groups
Arm/Group | Arm I (Docetaxel, Bintrafusp Alfa) | Arm II (Docetaxel) | Total
Number analyzed (Participants) | 6 | 3 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (7.44) | 69.0 (8.72) | 66.2 (7.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 4 | 3 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 3 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 3 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Smoking Status [Count of Participants; unit: Participants]
  Current | 0 | 1 | 1
  Former | 3 | 1 | 4
  Never | 3 | 1 | 4
MedDRA Disease Code [Count of Participants; unit: Participants]
  Lung adenocarcinoma | 6 | 0 | 6
  Squamous cell lung carcinoma | 0 | 1 | 1
  Non-small cell lung cancer, NOS | 0 | 2 | 2
ECOG Performance Status [Count of Participants; unit: Participants] — 0: Fully active, able to carry on all pre-disease performance without restriction>
  1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work> 0 is better than 1
  Participants
    0 | 4 | 1 | 5
    1 | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) of Bintrafusp Alfa in Combination With Docetaxel Versus (vs) Docetaxel Alone
Description: The primary analysis of PFS will be a comparison of the Kaplan-Meier curves for docetaxel + bintrafusp alfa vs. docetaxel alone using a one-sided log-rank test.
Time Frame: From randomization to the first of either disease progression or death from any cause, assessed up to 3 years and 2 months
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Arm I (Docetaxel, Bintrafusp Alfa): Patients receive docetaxel IV over 1 hour and bintrafusp alfa IV over 60 minutes on day 1. Treatment repeats every 3 weeks for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive bintrafusp alfa IV over 60 minutes on day 1. Cycles repeat every 3 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity. >
  * > >
  * > Bintrafusp Alfa: Given IV >
  * > >
  * > Docetaxel: Given IV
- Arm II (Docetaxel): Patients receive docetaxel IV over 1 hour on day 1. Cycles repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. Patients who experience disease progression may crossover to Arm I and receive bintrafusp alfa alone. >
  * > >
  * > Docetaxel: Given IV
Arm/Group | Arm I (Docetaxel, Bintrafusp Alfa) | Arm II (Docetaxel)
Number analyzed (Participants) | 6 | 3
months | 3.0 [1.7 to NA] — Not enough events to calculate an upper bound | 8.6 [1.8 to NA] — Not enough events to calculate an upper bound

2. Secondary Outcome: Overall Survival (OS)
Description: OS will be estimated using the Kaplan-Meier method, where the log-rank test will be used to compare the 2 treatment arms.
Time Frame: From study entry to death from any cause, assessed up to 3 years and 2 months
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Arm I (Docetaxel, Bintrafusp Alfa): Patients receive docetaxel IV over 1 hour and bintrafusp alfa IV over 60 minutes on day 1. Treatment repeats every 3 weeks for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive bintrafusp alfa IV over 60 minutes on day 1. Cycles repeat every 3 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity. >
  * > >
  * Bintrafusp Alfa: Given IV >
  * > >
  * Docetaxel: Given IV
- Arm II (Docetaxel): Patients receive docetaxel IV over 1 hour on day 1. Cycles repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. Patients who experience disease progression may crossover to Arm I and receive bintrafusp alfa alone. >
  * > >
  * Docetaxel: Given IV
Arm/Group | Arm I (Docetaxel, Bintrafusp Alfa) | Arm II (Docetaxel)
Number analyzed (Participants) | 6 | 3
months | 22.0 [6.3 to NA] — Not enough events to calculate an upper bound | 16.3 [1.8 to NA] — Not enough events to calculate an upper bound

3. Secondary Outcome: Confirmed Response Rates
Description: Will be classified as a confirmed response per the Immune-Modified Response Evaluation Criteria in Solid Tumors (iRECIST) criteria, if they have a partial or complete response for 2 consecutive evaluations at least 4 weeks apart. The proportion of patients with a confirmed response will be calculated and compared between the 2 arms using a Chi-square of Fisher's Exact test.
Time Frame: Up to 3 years and 2 months
Measure: Count of Participants; unit: Participants
Groups:
- Arm I (Docetaxel, Bintrafusp Alfa): Patients receive docetaxel IV over 1 hour and bintrafusp alfa IV over 60 minutes on day 1. Treatment repeats every 3 weeks for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive bintrafusp alfa IV over 60 minutes on day 1. Cycles repeat every 3 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity.
  >
  >
  >
  >
  >
  > Bintrafusp Alfa: Given IV
  >
  >
  >
  >
  >
  > Docetaxel: Given IV
- Arm II (Docetaxel): Patients receive docetaxel IV over 1 hour on day 1. Cycles repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. Patients who experience disease progression may crossover to Arm I and receive bintrafusp alfa alone.
  >
  >
  >
  >
  >
  > Docetaxel: Given IV
Arm/Group | Arm I (Docetaxel, Bintrafusp Alfa) | Arm II (Docetaxel)
Number analyzed (Participants) | 6 | 3
Participants | 1 | 0

4. Secondary Outcome: Duration of Response
Description: The duration of confirmed responses will be assessed using the Kaplan Meier method, where the duration of confirmed response will be defined as the time from the first documented date of response (complete response [CR] or partial response [PR]) to the date at which progression is first documented. Duration of response will be estimated using the Kaplan-Meier method, where the log-rank test will be used to compare the 2 treatment arms.
Time Frame: Up to 3 years and 2 months
Population: No confirmed response for Arm II.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Docetaxel, Bintrafusp Alfa) | Arm II (Docetaxel)
Number analyzed (Participants) | 1 | 0
months | 5.8 [5.8 to 5.8] |

5. Secondary Outcome: Incidence of Adverse Events
Description: The maximum grade for each type of adverse event will be summarized using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. The frequency and percentage of grade 3+ adverse events will be compared between the 2 treatment arms. Comparisons between arms will be made by using either the Chi-square or Fisher's Exact test.
Time Frame: Up to 3 years and 2 months
Population: Lower grades are better than higher grades
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Docetaxel, Bintrafusp Alfa) | Arm II (Docetaxel)
Number analyzed (Participants) | 6 | 3
Participants
  Grade 3+ Adverse Event | 3 | 3
  Grade 3+ Heme Adverse Event | 3 | 2
  Grade 3+ Non-Heme Adverse Event | 2 | 3
  Grade 4+ Adverse Event | 3 | 3
  Grade 4+ Heme Adverse Event | 3 | 2
  Grade 4+ Non-Heme Adverse Event | 0 | 1

ADVERSE EVENTS:
Time Frame: Up to 3 years and 2 months
Groups:
- Arm II Crossover (Docetaxel, Bintrafusp Alfa): Docetaxel: Given IV Docetaxel: Given IV
Arm/Group | Arm I (Docetaxel, Bintrafusp Alfa) | Arm II (Docetaxel) | Arm II Crossover (Docetaxel, Bintrafusp Alfa)
All-Cause Mortality (participants affected / at risk) | 0/6 | 1/3 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/3 | 0/1
Other Adverse Events (participants affected / at risk) | 3/6 | 1/3 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Docetaxel, Bintrafusp Alfa) (N=6) | Arm II (Docetaxel) (N=3) | Arm II Crossover (Docetaxel, Bintrafusp Alfa) (N=1)
Disease progression (General disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Docetaxel, Bintrafusp Alfa) (N=6) | Arm II (Docetaxel) (N=3) | Arm II Crossover (Docetaxel, Bintrafusp Alfa) (N=1)
Anemia (Blood and lymphatic system disorders) | 1 (5) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (5) | 0 (0) | 0 (0)
Fever (General disorders) | 2 (2) | 0 (0) | 0 (0)
Pain (General disorders) | 2 (3) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 0 (0) | 0 (0)
ECG QT corrected interval prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (2) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (3) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Weight loss (Investigations) | 1 (2) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 1 (3) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (3) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (5) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 1 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-25): https://cdn.clinicaltrials.gov/large-docs/35/NCT04396535/Prot_SAP_002.pdf
  • Informed Consent Form (2021-04-09): https://cdn.clinicaltrials.gov/large-docs/35/NCT04396535/ICF_001.pdf